CLINICAL TRIAL: NCT01346306
Title: Investigating Direct Current Stimulation as a Treatment for Depression: A Controlled Clinical Trial
Brief Title: Trial of Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC16360
Record Dates: First submitted 2011-04-13; First posted 2011-05-02 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCS 1 (Experimental)
  Interventions: Device: Eldith Company - direct current stimulator
- DCS 2 (Experimental)
  Interventions: Device: Eldith Company - direct current stimulator

INTERVENTIONS:
Device: Eldith Company - direct current stimulator — Direct current stimulation montage 1.
  Other Names: Neuroconn - direct current stimulator
  Arms: DCS 1
Device: Eldith Company - direct current stimulator — Direct current stimulation montage 2.
  Other Names: Neuroconn - direct current stimulator
  Arms: DCS 2

SUMMARY:
Among antidepressant treatments, ECT stands as the most effective in treating acute depression. However, patient concerns with the cognitive side effects of ECT have encouraged the development of new and more focal forms of brain stimulation such as transcranial Direct Current Stimulation (tDCS). However, not all patients may respond to this treatment in the way that it is currently administered and this has raised interest in finding alternative, possibly more optimal ways of administering tDCS. This study will investigate whether tDCS stimulation using an alternative electrode montage has antidepressant effects. Further sessions of tDCS, spaced less frequently, will be trialed for maintenance treatment. Mood, cognitive test performance and biomarkers will be measured periodically in the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets criteria for a DSM-IV Major Depressive Episode.
* Total MADRS score ≥20.

Exclusion Criteria:

* Diagnosis (as defined by DSM-IV) of: any psychotic disorder (lifetime); eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder (current or within the past year); mental retardation.
* History of drug or alcohol abuse or dependence (as per DSM-IV criteria) within the last 3 months (except nicotine and caffeine).
* Inadequate response to ECT in the current episode of depression.
* Subject is on regular benzodiazepine medication which it is not clinically appropriate to discontinue.
* Subject requires a rapid clinical response due to inanition, psychosis or high suicide risk.
* Neurological disorder or insult, e.g., recent stroke (CVA), which places subject at risk of seizure or neuronal damage with tDCS.
* Subject has metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
* Female subject who is pregnant.
* Participants who are not fluent in English will not be included in the trial for safety reasons: a) It is usually not possible to have an interpreter reliably available every weekday for up to 4 weeks and it is not safe to give tDCS to a subject who cannot tell us immediately of any side effects; b) As this is a novel treatment, the study involves detailed neuropsychological testing for safety reasons. This testing cannot be effectively or validly completed by someone who is not fluent in English. Note that translation of the proposed tests into English has not been validated and that we cannot be confident that neuropsychological impairment would be detected using this method.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, FRANZCP, MD, Principal Investigator — School of Psychiatry, University of New South Wales
Locations (2):
- Black Dog Institute, Randwick, New South Wales, Australia
- Singapore General Hospital, Singapore, Singapore